CLINICAL TRIAL: NCT07048691
Title: Prenatal and Postnatal Ultrasonographic Evaluation of Myelomeningocele to Predict Post-Surgical Outcomes
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHSW/Batch-Fall23/909
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Myelomeningocele
MeSH Terms: conditions — Meningomyelocele

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- G.E HEALTHCARE ultrasound machine with high-resolution convex probe
  Interventions: Diagnostic Test: G.E HEALTHCARE ultrasound machine with high-resolution convex probe

INTERVENTIONS:
Diagnostic Test: G.E HEALTHCARE ultrasound machine with high-resolution convex probe — After approval from the institutional ethical committee, a total number of patients presenting to the Radiology and Peads Neurosurgery department of Allied Hospital, Faisalabad, that met the inclusion criteria was selected. After obtaining informed consent from each patient and attendant of the patient, transabdominal ultrasound was examined longitudinal, transverse and oblique plans, ultrasound with a high- resolution convex probe was used by the radiologist

SUMMARY:
Myelomeningocele (MMC), also known as open spina bifida, is a serious congenital condition in which the cord and meninges protrude through the spinal column's defective bony encasement due to a defective closure of the posterior portion of the neural tube between the fourth week of pregnancy.

DETAILED DESCRIPTION:
The formation of the defect is influenced by both genetic and environmental factors, while the exact cause is yet unknown. There is currently no effective treatment for this common and debilitating central nervous system (CNS) dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 3rd trimester, Lesion between T1 and S1, Hindbrain herniation and Normal karyotype

Exclusion Criteria:

* Multiple gestation pregnancy
* Other fetal anomalies unrelated to myelomeningocele
* History of incompetent cervix, Other serious maternal medical conditions
* Inability to adhere to travel and follow-up requirements
* Contraindication to surgery and Inability to meet trial psychosocial criteria.

Ages: 28 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: After approval from the institutional ethical committee, a total number of patients presenting to the Radiology and Peads Neurosurgery department of Allied Hospital, Faisalabad, that met the inclusion criteria was selected. After obtaining informed consent from each patient and attendant of the patient, transabdominal ultrasound was examined longitudinal, transverse and oblique plans, ultrasound with a high- resolution convex probe was used by the radiologist.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
self administered questioner | 12 Months
  self administered questioner for yelomeningocele patients scroing range fron 0-40. 0 is for lower and 40 is worse and higher

CONTACTS AND LOCATIONS:
Locations (1):
- Allied Hospital, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No